CLINICAL TRIAL: NCT01209767
Title: Comparison of the Efficacy Between Cryolipolysis and Subcision for Treatment of Cellulite: A Prospective Randomized Control Trial.
Brief Title: Cryolipolysis and Subcision for Treatment of Cellulite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology - Head and Neck Surgery and Surgery-Organ Transplantation, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU34401
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Results first posted 2014-02-03 (Estimated); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Cellulite
Keywords: Cellulite; Cryolipolysis; Zeltiq; Subcision
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- cryolipolysis (Experimental)
  Interventions: Device: cryolipolysis
- subcision (Active Comparator)
  Interventions: Procedure: Subcision
- Control (Active Comparator): Areas with cellulite that had no treatment performed were considered the control arm.
  Interventions: Other: Control

INTERVENTIONS:
Device: cryolipolysis — During cryolipolysis, the system drew fat tissue into an applicator then exposed the extracted fat tissue to cold temperatures. The cold exposure caused fat cells to die, with the goal to decrease the raised areas of cellulite
  Arms: cryolipolysis
Procedure: Subcision — Subcision was performed by inserting a specially designed needle under the skin after local numbing medication is injected. The needle is moved in a repetitive motion parallel to the skin to separate the surface tissue from the deeper scar tissue with the goal to improve the dimpling caused by these tissues sticking together.
  Arms: subcision
Other: Control
  Other Names: No intervention in this group
  Arms: Control

SUMMARY:
This study intended to investigate and compare the changes that may occur in response to cryolipolysis (localized cool exposure) and subcision (surgical technique) on cellulite. The cryolipolysis cooling device used is FDA approved for skin cooling, but still investigational in the treatment of cellulite. It has previously been used for fat reduction on love handles or back fat. During cryolipolysis, the system drew fat tissue into an applicator then exposes the extracted fat tissue to cold temperatures. The cold exposure caused fat cells to die, with the goal to decrease the raised areas of cellulite. Subcision is a process used to treat scars left behind by acne or other skin diseases and has been noted to improve moderate to severe cellulite. Subcision is a simple surgical procedure that is performed by inserting a specially designed needle under the skin after local numbing medication is injected. The needle is moved in a repetitive motion parallel to the skin to separate the surface tissue from the deeper scar tissue with the goal to improve the dimpling caused by these tissues sticking together. This study was a pilot study designed to determine feasibility of these procedures.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female patients 18-60 years of age with more than one evident depressed lesion of cellulite on the upper thighs and/or buttocks.
* All subjects must have the affected areas that show the mattress phenomenon spontaneously when standing or while both lying and standing (Stage 2 or 3 of Nurnberger-Muller grading scale of cellulite7).
* Subjects who are willing and have the ability to understand and provide informed consent for participation in the study and are able to communicate with the investigator.

Exclusion Criteria:

* Pregnant or lactating
* Subjects who are unable to understand the protocol or to give informed consent.
* Subjects currently under treatment with an antiplatelet or anticoagulant for any medical problem or patients who have coagulation disorder.
* Subjects who have a known history of cold-induced disease such as cryoglobulinemia, paroxysmal cold hemoglobinuria, or cold urticaria.
* Subjects who have active skin disease or skin infection in treatment area.
* Subjects who are allergic to lidocaine or prilocaine.
* Subjects who are allergic to both cephalexin (and penicillin) AND levofloxacin (or another quinolone antibiotic).
* Subjects who have history of abnormal scarring.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2010-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects Receiving Split Body Treatment: The unit of randomization was the side of the body within each subject to receive either cryolipolysis or subcision.
  cryolipolysis : During cryolipolysis, the system drew fat tissue into an applicator and then exposed the extracted fat tissue to cold temperatures. The cold exposure caused fat cells to die, with the goal to decrease the raised areas of cellulite
  Subcision : Subcision was performed by inserting a specially designed needle under the skin after local numbing medication is injected. The needle was moved in a repetitive motion parallel to the skin to separate the surface tissue from the deeper scar tissue with the goal to improve the dimpling caused by these tissues sticking together.
Period: Overall Study
Arm/Group | Subjects Receiving Split Body Treatment
Started | 22
Completed | 18
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Subjects Receiving Split Body Treatment
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.4 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Blinded Rating of the Treatment Area (Cryolipolysis vs. Subcision) With the Best Cosmetic Appearance.
Description: Two dermatologists blindly evaluated and compared the treated and control areas of each side at the final follow up visit (week 12). They rated the area with the best cosmetic appearance and reported the percentages of participants for whom "Cryolipolysis" or "Subcision" resulted in the "best cosmetic appearance". It was possible for raters to determine that neither treatment outperformed the other, thereby rating the control arm better.
Time Frame: 12 weeks
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Groups:
- Cryolipolysis: cryolipolysis : During cryolipolysis, the system drew fat tissue into an applicator and then exposed the extracted fat tissue to cold temperatures. The cold exposure caused fat cells to die, with the goal to decrease the raised areas of cellulite
- Subcision: Subcision : Subcision was performed by inserting a specially designed needle under the skin after local numbing medication is injected. The needle is moved in a repetitive motion parallel to the skin to separate the surface tissue from the deeper scar tissue with the goal to improve the dimpling caused by these tissues sticking together.
- Control: Area that received no treatment
Arm/Group | Cryolipolysis | Subcision | Control
Number analyzed (Participants) | 18 | 18 | 18
Percentage of participants | 22.22 [6.41 to 47.64] | 33.33 [13.34 to 59.01] | 44.44 [21.53 to 69.24]

ADVERSE EVENTS:
Groups:
- Cryolipolysis: cryolipolysis : During cryolipolysis, the system drew fat tissue into an applicator then exposed the extracted fat tissue to cold temperatures. The cold exposure caused fat cells to die, with the goal to decrease the raised areas of cellulite
- Subcision: Subcision : Subcision was performed by inserting a specially designed needle under the skin after local numbing medication is injected. The needle was moved in a repetitive motion parallel to the skin to separate the surface tissue from the deeper scar tissue with the goal to improve the dimpling caused by these tissues sticking together.
- Control: Nothing was done to the area.
Arm/Group | Cryolipolysis | Subcision | Control
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 3/22 | 0/22
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cryolipolysis (N=22) | Subcision (N=22) | Control (N=22)
small ulcer (General disorders) | 0 (0) | 1 (1) | 0 (0)
lumps (General disorders) | 0 (0) | 2 | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes